CLINICAL TRIAL: NCT06552923
Title: Extension for Community Health Outcomes (ECHO) Diabetes Program
Acronym: ECHO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB201903243
Record Dates: First submitted 2024-08-08; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Federally Qualified Health Centers were randomized to start in 6-month phased entry and large, aggregate data for participating health centers was collected pre and post ECHO program
Masking Description: Masking was not used
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ECHO Intervention Immediate (Experimental): 9 FQHC were randomized to start the ECHO program June 2021. The providers at participating FQHCs joined tele-education one hour sessions and received CME for learning about diabetes care-related topics. They attended sessions twice monthly for 6-months
  Interventions: Other: ECHO Tele-Education
- ECHO Intervention Delayed (Experimental): 11 FQHC were randomized to start the ECHO program in December 2021. The providers at participating FQHCs joined tele-education one hour sessions and received CME for learning about diabetes care-related topics. They attended sessions twice monthly for 6-months
  Interventions: Other: ECHO Tele-Education

INTERVENTIONS:
Other: ECHO Tele-Education — A common curriculum was developed that covered best practices in multidisciplinary diabetes care for the primary care setting that was guided by the ADA Clinical Care. guidelines. FQHCs attended one-hour tele-ECHO sessions twice a month for 6-months.

SUMMARY:
The Project ECHO model is currently used in 180 countries to address chronic disease care through a provider empowerment, tele-education approach using a "hub" and "spoke" learning model. Few studies have rigorously evaluated the impact of the program on patient outcomes using randomized designs. This study evaluated implementation of an ECHO Diabetes program on patient-level, provider-level, and center-level outcomes in underserved populations receiving diabetes care from primary care providers.

Participants: Twenty Federally Qualified Health Centers (FQHCs) and FQHC "look alikes" across CA and FL were recruited to participate as spokes in the ECHO Diabetes trial. A stepped-wedge trial design was used with randomized, phased-in intervention entry for participating health centers (or "spokes").

Interventions: Spokes were provided access to 6-months of tele-education sessions with continuing medical education credits, access to real-time support for complex medical decision making with hub subspecialty teams, and access to a diabetes support coach.

Main outcomes and Measures: Participating FQHCs ("spokes") provided aggregate data including Healthcare Effectiveness Data and Information Set (HEDIS) reporting on the % of patients with HbA1c >9%.

DETAILED DESCRIPTION:
The recruitment of spokes for the ECHO Diabetes program was accomplished by focusing on FQHC (and FQHC look-alikes) through use of the Neighborhood Deprivation Index coupled with provider geocoding. This novel approach ensured recruitment of spokes that deliver care for communities in medically underserved areas. Over 30 million people in the U.S. receive primary care in FQHCs. Federal funding requirements for FQHCs mandate that no one is turned away for care based on insurance status, that need-based sliding scales are used for payment, and that the healthcare providers must be representative of the communities they serve (i.e., language needs, race, and ethnicity).

Any healthcare provider from the participating spoke sites were eligible for the ECHO Diabetes intervention. Healthcare providers at participating spokes were offered the opportunity to attend real-time, interactive, one-hour, bimonthly, tele-education sessions with continuing medical education credits provided. The curriculum was designed using the current standards of diabetes care and delivered by a team of multidisciplinary experts including adult endocrinologists, pediatric endocrinologists, clinical health psychologists, exercise physiologists, pharmacists, diabetes education and care specialists (CDCES), registered dietitians, and medical sociologists. Each tele-ECHO Diabetes session was recorded and available on-demand for healthcare providers at participating spoke sites, along with access to an online repository of diabetes resources and guidelines. Providers were also able to reach out to the hub team for real-time support with complex medical decision making, as needed. Finally, spokes also had access to Diabetes Support Coaches for their patients. A full description of the use of Diabetes Support Coaches in the ECHO Diabetes program has been published elsewhere and involved using a combination of a community health worker (CHW) and peer mentors to address social determinants of health (SDOH), and to create more community capacity within the spokes for people with diabetes.

ECHO Diabetes utilized a variation of a stepped-wedge study design, allowing for two phases of program kick-off and patient recruitment at spokes. Spoke sites provided basic metrics of their patient panels, including the number of clinic locations participating in the program, and adults with T1D and T2D. Covariate-constrained randomization was used to assign spokes to begin the ECHO Diabetes intervention in May or December of 2021. The randomization design specifications allowed for clinic arm totals to differ by no more than one, and the mean number of patients with diabetes to not differ by greater than 20% between arms. Final randomized intervention assignment was distributed to enrolled spokes in Spring of 2021. Spoke-level data capture incorporated the transfer of aggregate-level data by participating centers for calendar years 2020, 2021, 2022 including Health Effectiveness Data and Information Set (HEDIS) and Uniform Data System (UDS) diabetes-related measures.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Seen for routine care at participating FQHC
* Diagnosis of Type 1 Diabetes or Type 2 Diabetes

Exclusion Criteria:

• Not meeting all inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32796 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
HbA1c | 6-months
  The percent of patients with HbA1c greater than 9 percent

CONTACTS AND LOCATIONS:
Overall Officials: David Maahs, PhD, MD, Principal Investigator — Stanford University; Michael Haller, MD, Principal Investigator — University of Florida; Ashby F Walker, PhD, Principal Investigator — University of Florida
Locations (17):
- United States (17):
  - CommuniCare Davis Family Health Center, Davis, California
  - St Agnes Medical Center, Fresno, California
  - La Clinica, Multiple Locations, California
  - Santa Rosa Community Health Centers, Multiple Locations, California
  - Shasta Community Health Centers, Multiple Locations, California
  - Health Service Alliance, Rancho Cucamonga, California
  - Hill Country Community Clinic, Redding, California
  - CommuniCare Salud Family Health, West Sacramento, California
  - CommuniCare Hansen Family Center, Woodland, California
  - Premier Community Health, Dade City, Florida
  - Community Health of South Florida (CHI), Homestead, Florida
  - Banyan Health Systems, Miami, Florida
  - Borinquen Medical Center, Miami, Florida
  - Orange Blossom Family Health, Orlando, Florida
  - Evara Health System, Pinellas Park, Florida
  - Tampa Family Health Center, Tampa, Florida
  - Treasure Coast Community Health, Vero Beach, Florida

IPD SHARING:
Plan to Share IPD: No